CLINICAL TRIAL: NCT06358885
Title: IGHID 12230 - Scaling up the Brief Alcohol Intervention to Prevent HIV Infection in Vietnam: a Cluster Randomized, Implementation Trial (EBAI)
Brief Title: IGHID 12230 - An Implementation Trial of an Experiential Brief Alcohol Intervention for HIV Prevention
Acronym: EBAI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institutes of Health (NIH) (NIH); Hanoi Medical University (Other); Johns Hopkins University (Other); University of Washington (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 22-3123; R01AA030480 (NIH)
Record Dates: First submitted 2024-04-01; First posted 2024-04-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-06

CONDITIONS: HIV-1-infection; Unhealthy Alcohol Use
Keywords: Alcohol intervention; Cluster randomized controlled implementation trial; Implementation Science; HIV/AIDS; Antiretroviral therapy; Cognitive behavioral therapy; Motivational Interviewing; Motivational Enhancement Therapy; Cost Analysis; Economic Evaluation; Vietnam
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: A two-arm cluster-randomized implementation trial comparing two strategies to scale-up an evidence-based brief alcohol intervention (BAI), in Vietnam, examining the mechanisms of BAI scale-up and the impact of experiential BAI (EBAI) on clinic staff. The two implementation approaches are facilitation only (FAC) and facilitation plus an experiential brief alcohol intervention (EBAI+FAC).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitation Only (FAC) (Active Comparator): Clinics randomized to the FAC arm will implement BAI delivery to PWH using the facilitation only approach.
  Interventions: Other: Facilitation (FAC)
- Facilitation Plus an Experiential Brief Alcohol Intervention (EBAI+FAC) (Experimental): Clinics randomized to the EBAI+FAC arm will implement BAI delivery to PWH participants using the facilitation approach. Additionally, clinic staff, irrespective of their own alcohol use, will be offered the BAI themselves prior to delivering the BAI.
  Interventions: Other: Facilitation (FAC); Behavioral: Experiential Brief Alcohol Intervention (EBAI)

INTERVENTIONS:
Other: Facilitation (FAC) — The facilitation approach will use a flexible clinic level implementation strategy that helps clinics to address common barriers, such as counselor skills, competing priorities, and resource deficits.
Behavioral: Experiential Brief Alcohol Intervention (EBAI) — Clinic staff will be offered the experiential BAI prior to implementation. The BAI comprises 2 in-person sessions and 2 booster phone sessions. Clinic staff responsible for delivering the BAI to PWH participants will be offered 3 additional consolidation sessions to integrate their experiences receiving the BAI with their delivery of the BAI.
  Arms: Facilitation Plus an Experiential Brief Alcohol Intervention (EBAI+FAC)

SUMMARY:
This study is a hybrid type 3, cluster randomized implementation trial to examine effective strategies to scale up the Brief Alcohol Intervention (BAI) in ART clinics in Vietnam. One arm will receive only facilitation for BAI implementation. Facilitation is a flexible strategy that helps clinics to address common barriers, such as counselor skills, competing priorities, and resource deficits. In the other arm, in addition to facilitation, clinic staff, irrespective of their own alcohol use, will be offered the BAI themselves as experiential learning (EBAI) to address their own alcohol-related attitudes and behaviors. Clinic staff responsible for delivering the BAI to patients will also be offered 3 consolidation activities to integrate their own experiences with their delivery of the BAI.

DETAILED DESCRIPTION:
In this cluster-randomized controlled, hybrid type 3 implementation trial, investigators will assess two approaches to the brief alcohol intervention (BAI) scale-up. The BAI is an evidence-based intervention to address unhealthy alcohol use that comprises 2 in-person sessions and 2 booster telephone sessions. Face-to-face 45-minute sessions occur ~1 month apart; 10-minute telephone sessions occur 2 to 3 weeks after each face-to-face session. Investigators chose a hybrid type 3 design to evaluate implementation outcomes, while simultaneously ensuring that effectiveness outcomes, specifically viral suppression, are achieved. Investigators will compare facilitation (FAC) versus EBAI+FAC in 30 ART clinics in Vietnam. The FAC arm, the comparison arm, will use internal and external facilitators to help clinics and staff address common barriers to BAI implementation. Facilitation typically works through interactive problem solving and support. In the EBAI+FAC arm, clinic staff, defined as clinic directors, physicians, nurses, and counselors, will be offered the experiential BAI (EBAI), regardless of their own alcohol use, prior to BAI implementation, and clinic staff responsible for delivering the BAI to patients will also be offered 3 additional consolidation opportunities to integrate their own experiences with their delivery of the BAI to PWH. Randomization will be 1:1 with 15 clinics per arm. Clinics will be assessed pre-training for key contextual factors, related to clinic characteristics and clinic staff.

Upon trial initiation, persons with HIV (PWH) initiating or on ART will be screened for unhealthy alcohol use with the AUDIT-C (Time 0). Those PWH who screen positive for unhealthy alcohol use will be offered the BAI by trained clinic counselors. PWH who do not screen positive will continue to be screened with the AUDIT-C at routine ART clinic visits. PWH who screen positive but refuse to participate in the trial or are excluded due to alcohol withdrawal symptoms will continue to be screened with the AUDIT-C at every routine ART clinic visit per standard clinic procedures. PWH may decline AUDIT screening when it is offered. Implementation and effectiveness outcomes will be evaluated to 12 or 24 months (Aim 1). After the 12- month assessments, mechanisms underlying successful implementation in both arms will be explored using qualitative and quantitative methods (Aim 2). Investigators will explore the effect of implementing the BAI (both arms) and experiencing the BAI (EBAI+FAC arm) on staff members' alcohol use and attitudes toward alcohol and BAI (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

PWH cohort participants

* Person living with HIV at any stage of HIV infection
* Currently attending the study ART clinic at any ART stage (initiating or receiving ART)
* AUDIT-C score >=4 for men or >=3 for women
* >= 18 years of age
* Willing to provide informed consent, which includes consenting to interview and collection of dried blood spots

Clinic staff participants:

* Work at the ART clinic as a clinic director, physician, nurse, or counselor
* Willing to provide informed consent

Exclusion Criteria:

PWH cohort participants:

* Psychological disturbance preventing participation
* Cognitive impairment
* Threatening behavior
* Unwilling to provide locator information Note: If a participant screens positive with the AUDIT-C and is identified to be at substantial risk for alcohol withdrawal based on the Mini International Neuropsychiatric Interview (MINI) and Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA) will be referred for treatment. They will not be eligible for enrollment until after alcohol withdrawal concerns are addressed.
* These participants may be rescreened, consented, and enrolled after treatment.

Clinic staff participants:

* Psychological disturbance, cognitive impairment, or threatening behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3234 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Fidelity Score | 15 months
  Fidelity is a clinic-level measure assessed as a composite of the recipients of the BAI. The timeframe of 15 months reflects individual recruitment over 12 months plus 3 months for completion of the BAI.
  The score comprises successful completion of the 4 protocol-specified BAI sessions (2 in-person, 2 by phone) within 7 weeks of the initial session weighted by the central fidelity rater's quality rating of the in-person sessions. Fidelity will be assessed using a tailored selection of fidelity measures including the BAI Core Components Checklist. The clinic fidelity score ranges from 0-100. The score will be the percentage of counseling sessions completed, multiplied (weighted) by the combined average quality rating of counseling sessions. Higher scores indicate higher fidelity.
Viral Suppression | 12 months
  Viral suppression is defined as a viral load <1000 copies/mL on a dried blood spot (DBS) sample collected 12 months after enrollment of a participant.

SECONDARY OUTCOMES:
BAI Acceptability Score - Clinic Staff: Acceptability of Intervention Measure (AIM) scale | Up to 12 months
  Acceptability is the perception that the BAI intervention is agreeable, palatable, or satisfactory to clinic staff.
  Acceptability among clinic staff will be assessed using the Acceptability of Intervention Measure (AIM), which consists of 4 items containing responses on a 5-point Likert scale, ranging from 1-4.
  The AIM score will be the mean of the 4 item responses (range: 1-5). Higher AIM scores indicate higher acceptability.
BAI Acceptability score Counselors: Mental Health Implementation Science Tools (mhIST) Acceptability Scale for Providers | Up to 12 months
  Acceptability is the perception that the BAI intervention is agreeable, palatable, or satisfactory to counselors delivering the BAI to patients.
  Acceptability among counselor participants will be assessed using the Mental Health Implementation Science Tools (mhIST) Acceptability Scale for providers, which consists of 13 items containing responses on a 4-point Likert scale, ranging from 0-3. The mhIST score is calculated as the mean score of all responses (range: 0-39). Higher mhIST scores indicate higher acceptability.
BAI Acceptability PWH: Mental Health Implementation Science Tools (mhIST) Acceptability Scale for Consumers | Up to 12 months
  Acceptability is the perception that the BAI intervention is agreeable, palatable, or satisfactory to PWH.
  Acceptability among PWH participants will be assessed using the Mental Health Implementation Science Tools (mhIST) Acceptability Scale for consumers, which consists of 15 items containing responses on a 4-point Likert scale ranging from 0-3. The mhIST score is calculated as the mean score of all responses (range: 0-45). Higher mhIST scores indicate higher acceptability.
Penetration- Proportion of PWH Screened with the AUDIT-C | Up to 12 months
  The first penetration metric will be the: proportion of PWH initiating or on ART who are screened with the AUDIT-C.
Penetration - Proportion of PWH who screen positive who receive at least one counseling session | Up to 12 months
  The second penetration metric will be the proportion of PWH that screen positive who receive at least one BAI counseling session.
Costs | Up to 24 months
  Investigators will use an "ingredients" or bottom-up approach, with comparison to "top-down" costing. The cost estimates will follow the investigators published conceptual framework for assessing implementation costs and cost analysis of health services. Investigators will include all types of measurable costs (e.g., staff, equipment, consumables, overheads, etc.) associated with key steps and component of the respective implementation strategy and BAI service delivery. Investigators will follow international conventions for all procedures including economic costing, discounting, and reporting.
Sustainability Score: Provider Support of Sustainment Scale (PRESS) | Up to 24 months
  Sustainability will be measured among clinic staff, including directors, using the provider support of sustainment scale (PRESS), a brief, 3-item measure of sustainment that is pragmatic and useable across different evidence-based intervention (EBIs), provider types, and settings. Responses are recorded on a 5-point scale ranging from 0 (not at all) to 4 (to a very great extent) and the score is calculated as the mean of the 3 responses with higher scores indicating higher sustainability. The PRESS captures frontline staff's report of their clinic's continued use of an EBI.
AUDIT (total score) - Clinic staff | Up to 24 months
  Investigators will assess the total Alcohol Use Disorders Identification Test (AUDIT) score. The AUDIT is a 10-item scale with summed responses ranging from 0-40; higher scores indicating more harmful alcohol consumption.
AUDIT (total score) - PWH | Up to 12 months
  Investigators will assess the total Alcohol Use Disorders Identification Test (AUDIT) score. The AUDIT is a 10-item scale with summed responses ranging from 0-40; higher scores indicating more harmful alcohol consumption.
Fidelity (Extended Window) | 17 months
  Fidelity is a clinic-level measure assessed as a composite of the recipients of the BAI. The timeframe of 17 months reflects individual recruitment over 12 months plus 5 months for completion of the BAI.
  The score comprises successful completion of the 4 protocol-specified BAI sessions (2 in-person, 2 by phone) within 4 months of the initial session weighted by the central fidelity rater's quality rating of the in-person sessions. Fidelity will be assessed using a tailored selection of fidelity measures including the BAI Core Components Checklist. The clinic fidelity score ranges from 0-100. The score will be the percentage of counseling sessions completed, multiplied (weighted) by the combined average quality rating of counseling sessions. Higher scores indicate higher fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Go, MD, Principal Investigator — University of North Carolina
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator who proposes to use the data has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Bartels SM, Phan HTT, Hutton HE, Nhan DT, Sripaipan T, Chen JS, Rossi SL, Ferguson O, Nong HTT, Nguyen NTK, Giang LM, Bui HTM, Chander G, Sohn H, Kim S, Tran HV, Nguyen MX, Powell BJ, Pence BW, Miller WC, Go VF. Scaling up a brief alcohol intervention to prevent HIV infection in Vietnam: a cluster randomized, implementation trial. Implement Sci. 2024 Jun 12;19(1):40. doi: 10.1186/s13012-024-01368-6. PMID 38867283

DOCUMENTS (1):
  • Informed Consent Form (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT06358885/ICF_000.pdf